CLINICAL TRIAL: NCT05799547
Title: The Effect of Cold Application on the Pain, Comfort and Satisfaction of the Patient on First Standing After Cesarean Section
Brief Title: The Effect of Cold Application on Patient's Pain, Comfort and Satisfaction After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 55555
Record Dates: First submitted 2023-01-10; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- experimental group (Experimental)
  Interventions: Other: cold group

INTERVENTIONS:
Other: cold group — Application will be made in the form of 10 minutes of application to the cesarean section incision, 20 minutes of break and 10 minutes of application.
  Arms: experimental group

SUMMARY:
A healthy postpartum period is important for the health of the mother and baby. One of the main problems that occur after cesarean section, which is a major surgical procedure, is pain. However, since the mother is in the postpartum period, she may have problems in her own care, healing process and baby care due to pain. Non-pharmacological treatment is methods such as massage, acupressure, hot and cold application that can be applied at birth to support scientific medicine. The cold application examined in our research, is among these applications. participants will be determined by the block randomization method. Cold application will be applied to the cesarean section site of the patient for 10 minutes in the experimental group, followed by a break of 20 minutes, followed by a 10-minute application, and immediately after the application, the patient will stand up. Only the routine practice of the clinic will be applied to the control group. Data; will be collected using the introductory information form, visual analog scale (VAS) and cold application satisfaction evaluation form. When the studies were examined, no other study was found in the same application as our study. Therefore, in this study, it was aimed to evaluate the effect of cold application on the patient's pain during the first leg, the need for painkillers and satisfaction, due to the higher first take-off pain after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women who had cesarean section surgery
* Having had a previous cesarean section,

Exclusion Criteria:

* Those who have problems in postpartum vital signs and bleeding control
* Those who have systemic diseases that may affect cold application
* Those who are distressed and not suitable for practice by the service midwives and doctors,
* Those who do not want to participate in the research

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-07-10 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) | 1 week
  The visual analog scale is used to assess pain. The person marks the pain he feels on a ten-centimeter chart that expresses the absence of pain on one side and the pain he feels at the peak on the other side.